CLINICAL TRIAL: NCT04128566
Title: MechSens - Dose-response Relationship of in Vivo Ambulatory Load and Mechanosensitive Cartilage Biomarkers: the Role of Age and Tissue Health
Brief Title: MechSens - Dose-response Relationship of in Vivo Ambulatory Load and Mechanosensitive Cartilage Biomarkers
Acronym: MechSens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-01315;ch19Muendermann3
Record Dates: First submitted 2019-10-03; First posted 2019-10-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Articular Cartilage Degeneration
Keywords: articular cartilage; mechanosensitive blood markers of articular cartilage; walking stress test; ambulatory load; articular cartilage thinning; anterior cruciate ligament (ACL) injury; articular cartilage quality
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Masking Description: Blinding to the experimental condition is not possible because of the obvious differences between conditions (partial weight bearing and additional load). However, the person processing the data will be blinded to the condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: healthy subjects aged between 20 and 30 years (Experimental): healthy subjects aged between 20 and 30 years
  Interventions: Procedure: walking stress test
- Group 2: previous ACL injury aged between 20 and 30 years (Experimental): subjects with previous Anterior cruciate Ligament (ACL) injury aged between 20 and 30 years
  Interventions: Procedure: walking stress test
- Group 3: healthy subjects aged between 40 and 60 years (Experimental): healthy subjects aged between 40 and 60 years
  Interventions: Procedure: walking stress test
- previous ACL injury aged between 40 and 60 years (Experimental): subjects with previous ACL injury aged between 40 and 60 years
  Interventions: Procedure: walking stress test

INTERVENTIONS:
Procedure: walking stress test — walk for 30 minutes on a treadmill with either one of the three loading conditions (reduced load = 80% Bodyweight (BW), normal load = 100% BW, increased load = 120% BW). The order of experimental condition will be applied in randomized order determined by block randomization, and the same self-selected walking speed will be used for all conditions.

SUMMARY:
This study is to investigate the effects of age, tissue status and the presence of inflammation on the in vivo dose-response relationship of ambulatory load and mechanosensitive blood markers of articular cartilage.

DETAILED DESCRIPTION:
Articular cartilage is an avascular and aneural tissue that facilitates joint motion with minimal friction. Osteoarthritis (OA) is a joint disease that affects the whole joint resulting in severe articular cartilage degeneration with a prevalence worldwide of more than 10%. Although the molecular mechanisms that trigger the pathological changes in OA are largely unknown, the ability of chondrocytes to respond to load is believed to play a critical role in maintaining healthy tissue and in the initiation of OA. Different modes of ambulation have resulted in increases of specific blood markers, and immobilization during bed-rest lead to reductions in the same blood markers. However, the dose-response relationship between ambulatory load and mechanosensitive blood markers, its biological variation in healthy persons and in patients with a high risk of developing OA (e.g. with increasing age or after joint injury), and its relevance for cartilage degeneration are unknown. Based on reported differences in the magnitude of load-induced changes in blood markers of articular cartilage depending on the type of physical activity,an experimental framework of a systematic and controlled modulation of weight bearing during a walking stress test was previously tested and will be employed in this study. The following specific aims will be addressed:

Specific Aim 1: Investigate the in vivo dose-response relationship between ambulatory load and mechanosensitive blood markers of articular cartilage using controlled weight bearing during a walking stress test and age, tissue status and the presence of inflammation as experimental paradigms.

Specific Aim 2: Investigate the prognostic ability of the individual in vivo dose-response relationship between ambulatory load and mechanosensitive blood markers of articular cartilage for articular cartilage degeneration.

Healthy subjects and subjects with previous anterior cruciate ligament (ACL) injury aged 20 to 50 years will be clinically assessed, undergo magnetic resonance imaging (MRI) of both knees, and complete questionnaires on physical function and physical activity. Participants will wear an activity monitor for the 7 days before and during the experiment to record their physical activity level. Each participant will complete three walking stress tests (30 minutes walking) on separate days with repeated blood sampling to assess load-induced changes in levels of mechanosensitive blood markers (COMP, MMP-3, PRG-4, ADAMTS-4). In each test, one of three different ambulatory loads will be applied (80, 100 and 120% body weight (BW)). Inflammation will be assessed as IL-6 serum concentration. Tissue status of articular knee cartilage will be assessed as MRI T2 relaxation time and cartilage thickness at baseline and at 24-month follow-up.

ELIGIBILITY:
Inclusion Criteria for group 1 and 3:

* Being physically active (>2hours/week)
* No previous known knee injury:

Inclusion Criteria for group 2 and 4:

* Being physically active (>2hours/week)
* ACL rupture between 2 to 10 years prior to the study

Exclusion Criteria:

* Inability to provide informed consent
* Age < 20 years (before maturation) or age > 60 years
* Advanced general sarcopenia (degenerative loss of muscle mass in aging) and high likelihood of osteoarthritic changes
* Body mass index (BMI) > 35 kg/m2:
* Excessive skin movement that influences the gait analysis
* Inability to walk for 30 minutes
* Contraindications for a knee MRI
* Active rheumatic disorder
* Prior neuromuscular impairment (e.g. stroke)
* Conditions other than knee injury that could cause abnormal patterns of locomotion
* Prior hip, knee, and ankle prosthesis
* Osteotomy of the lower extremities - Prior spine surgery
* Other major medical problems
* Pregnancy
* Investigators and their immediate families are not permitted to be subjects
* Persons who have previously completed or withdrawn from this study
* Patients currently enrolled in another experimental (interventional) protocol

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Change in serum levels of Interleukin 6 (IL-6), ( mechanosensitive blood marker of articular cartilage) in pg/ml | Before walking stress test (t0= Baseline), immediately after walking stress test (t1), 30-minutes after walking stress test (t2) and after two additional 90-minute resting intervals after walking stress test (t3 and t4)
  Change in serum level of Interleukin 6 (IL-6), (mechanosensitive blood marker of articular cartilage) in pg/ml
Change in serum levels of Cartilage oligomeric matrix Protein (COMP) (mechanosensitive blood marker of articular cartilage) in U/l | Before walking stress test (t0= Baseline), immediately after walking stress test (t1), 30-minutes after walking stress test (t2) and after two additional 90-minute resting intervals after walking stress test (t3 and t4)
  Change in serum levels of Cartilage oligomeric matrix Protein (COMP) (mechanosensitive blood marker of articular cartilage) in U/l
Change in serum levels of Matrix metallopeptidase (MMP)-3 (mechanosensitive blood marker of articular cartilage) in ng/ml | Before walking stress test (t0= Baseline), immediately after walking stress test (t1), 30-minutes after walking stress test (t2) and after two additional 90-minute resting intervals after walking stress test (t3 and t4)
  Change in serum levels of Matrix metallopeptidase (MMP)-3 (mechanosensitive blood marker of articular cartilage) in ng/ml
Change in serum levels of Matrix metallopeptidase (MMP)-9 (mechanosensitive blood marker of articular cartilage) in ng/ml | Before walking stress test (t0= Baseline), immediately after walking stress test (t1), 30-minutes after walking stress test (t2) and after two additional 90-minute resting intervals after walking stress test (t3 and t4)
  Change in serum levels of Matrix metallopeptidase (MMP)-9 (mechanosensitive blood marker of articular cartilage) in ng/ml
Change in serum levels of Proteoglycan (PGR)-4 (mechanosensitive blood marker of articular cartilage) in mg/ml | Before walking stress test (t0= Baseline), immediately after walking stress test (t1), 30-minutes after walking stress test (t2) and after two additional 90-minute resting intervals after walking stress test (t3 and t4)
  Change in serum levels of Proteoglycan (PGR)-4 (mechanosensitive blood marker of articular cartilage) in mg/ml
Change in serum levels of A disintegrin and metalloproteinase with thrombospondin motifs (ADAMTS-4) (mechanosensitive blood marker of articular cartilage) in ng/mL | Before walking stress test (t0= Baseline), immediately after walking stress test (t1), 30-minutes after walking stress test (t2) and after two additional 90-minute resting intervals after walking stress test (t3 and t4)
  Change in serum levels of A disintegrin and metalloproteinase with thrombospondin motifs (ADAMTS-4) (mechanosensitive blood marker of articular cartilage) in ng/mL

SECONDARY OUTCOMES:
Change in modified Knee Society Score (KSS) score | Before walking stress test (t0= Baseline), at 12-month follow-up, at 24-month follow-up
  KSS consists of a total of 34 questions divided into four subscales which are rated separately. It consists of a Knee Score, which only rates the knee joint itself (e.g. pain, range of motion, stability and radiographic alignment), and a Function Score (patient's walking distance, climbing stairs and use of walking aids). The higher the score, the better the outcome in all subscales.
Change in modified Knee Injury and Osteoarthritis Outcome Score (KOOS) score | Before walking stress test (t0= Baseline), at 12-month follow-up, at 24-month follow-up
  The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). The five KOOS subscales rate on a 5-point Likert-scale as extremely important, very important, moderately important, somewhat important, or not important at all.
Change in Physical activity (PA) level | during the 7 days prior to Baseline and during the Walking stress test (t0= Baseline)
  PA level ( number of steps taken, PA intensity) will be recorded using an activity monitor (ActiGraph GT3X+, Pensacola, FL, USA)
Joint kinematics and kinetics | during the Walking stress test (t0= Baseline)
  For the the three loading conditions at the Walking stress test, an inertial sensor system (RehaGait®, Hasomed GmbH, Magdeburg, Germany) will be used to collect joint angle curves at the ankle, knee and hip.
Change in heart rate (beats per minute) | During the walking stress test until 10 minutes after the stress test
  To assess and compare the cardiovascular stress subjects experience during the walking stress tests the heart rate will be measured.
Change in T2 relaxation time from baseline to follow-up | MRI at least 7 days prior to the Walking stress test (t0= Baseline) and MRI 24 months after baseline
  Tissue status will be determined by the T2 relaxation time of weight bearing knee cartilage analyzed by Magnetic resonance Imaging (MRI) of both knees
Change in cartilage thickness from baseline to follow-up | MRI at least 7 days prior to the Walking stress test (t0= Baseline) and MRI 24 months after baseline
  Tissue status will be determined by the thickness of weight bearing knee cartilage analyzed by Magnetic resonance Imaging (MRI) of both knees

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Muendermann, Prof. Dr., Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Kunzler M, Herger S, De Pieri E, Egloff C, Mundermann A, Nuesch C. Effect of load carriage on joint kinematics, vertical ground reaction force and muscle activity: Treadmill versus overground walking. Gait Posture. 2023 Jul;104:1-8. doi: 10.1016/j.gaitpost.2023.05.018. Epub 2023 May 19. PMID 37263066
- [Derived] Herger S, Vach W, Nuesch C, Liphardt AM, Egloff C, Mundermann A. Dose-response relationship of in vivo ambulatory load and mechanosensitive cartilage biomarkers-The role of age, tissue health and inflammation: A study protocol. PLoS One. 2022 Aug 19;17(8):e0272694. doi: 10.1371/journal.pone.0272694. eCollection 2022. PMID 35984848